CLINICAL TRIAL: NCT01444196
Title: Multi-center, Double Blind, Dose Escalating Study to Compare the Effects of 5 mg, 10mg and 20mg of Desloratadine in Patients With Acquired Cold Urticaria (ACU)
Brief Title: Desloratadine 5, 10 and 20mg in Patients With Cold Urticaria
Acronym: AECUDATT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marcus Maurer (Other)
Collaborators: Johannes Gutenberg University Mainz (Other)
Responsible Party: Sponsor-Investigator, Marcus Maurer, Head of Research Dept. of Dermatology, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-005746-22; 2008-005746-22 (EudraCT Number)
Record Dates: First submitted 2011-09-29; First posted 2011-09-30 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Urticaria
Keywords: ACU; acquired cold urticaria
MeSH Terms: conditions — Urticaria | interventions — desloratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desloratadine dose (Other): 1. Study group: 5 mg Desloratadine during the whole study
  2. Study group: 5 mg every day for 14 (+-2 days) start with Visit 2, 10 mg every day for 14 (+-2 days) start with Visit 3, 20 mg every day for 14 (+-2 days) start with Visit 4.
  Interventions: Drug: Desloratadine
- Dose of Desloratadine (Other): 1. Study group: 5 mg Desloratadine during the whole study
  2. Study group: 5 mg every day for 14 (+-2 days) start with Visit 2, 10 mg every day for 14 (+-2 days) start with Visit 3, 20 mg every day for 14 (+-2 days) start with Visit 4.
  Interventions: Drug: Desloratadine

INTERVENTIONS:
Drug: Desloratadine — Every day,per mouth,in the evening, for 14 +- 2 days.
  Other Names: No arm names.

SUMMARY:
The primary objective of the study is to assess the dosis of DL which is sufficient to inhibit cold urticaria symptoms.

DETAILED DESCRIPTION:
A total of 30 patients (male and female) with ACU will be included in this study

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated
* Reliable method of contraception for both women of childbearing potential as well as man during the study and 3 months thereafter. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner
* Outpatients with ACU for more than 6 weeks. Urticaria symptoms must comprise wheal and itch.
* Age between 18 and 75 years

Exclusion Criteria:

* Subjects who are inmates of psychiatric wards, prisons, or other state institutions. Existing or planned placement in an institution after ruling according to § 40 passage 1 number 4 AMG (Arzneimittelgesetz).
* The presence of permanent severe diseases, especially those affecting the immune system, except urticaria and cold urticaria
* The presence of permanent gastrointestinal condition which may influence the oral therapy (chronic diarrhoea diseases, congenital malformations or surgical mutilations of gastrointestinal tract)
* History or presence of epilepsy, significant neurological disorders, cerebrovascular attacks or ischemia
* History or presence of myocardial infarction or cardiac arrhythmia which requires drug therapy
* Evidence of severe renal dysfunction
* Evidence of significant hepatic disease (liver enzymes twice the upper reference value)
* History of adverse reactions to DL
* Presence of active cancer which requires chemotherapy or radiation therapy
* Presence of alcohol abuse or drug addiction
* Intake of oral corticosteroids within 14 days prior to screening visit
* Use of depot corticosteroids or chronic systemic corticosteroids within 21 days prior to screening visit
* Use of systemic immunosupressants/immunomodulators like ciclosporine A, dapsone, methotrexate, mycophenolate, chloroquine, and comparable drugs within 28 days prior to screening visit.
* Pregnancy or breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
CTTs and CSTTs assessed by TEMPtest 3.0 + urticaria network SOPs | 6 weeks

SECONDARY OUTCOMES:
Presence of wheal(s) at 4°C Intensity of pruritus and burning Number and duration of angioedemas QoL as assessed by DLQI Severity of ACU (by ACUSI) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Maurer, Prof., Principal Investigator — Charite, University
Locations (1):
- Department of Dermatology, Venerology and Allergology, Berlin, State of Berlin, Germany

REFERENCES:
- See also: Kälteurtikaria — http://urtikaria.net